CLINICAL TRIAL: NCT03023072
Title: Evaluation of an Incontinence Product
Status: Terminated | Type: Observational
Why Stopped: Site no longer met criteria
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-CWS2016-001
Record Dates: First submitted 2017-01-12; First posted 2017-01-18 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Phase 1: Subjects will use the incontinence pad with incontinence detection notifications turned on
  Interventions: Other: Incontinence Detection System
- Phase 2: Subjects will use the incontinence pad with incontinence notification turned off

INTERVENTIONS:
Other: Incontinence Detection System
  Groups: Phase 1

SUMMARY:
The purpose of this study is to determine if the sponsor's Incontinence Product reduces patient exposure time to a wet and/or soiled incontinence pad.

ELIGIBILITY:
Inclusion Criteria:

* English speaking/reading adults, age ≥ 18 years
* Incontinent (fecal, urine, or dual incontinence)
* Patients with dual incontinence who require use of a fecal management system (but no urinary catheter)
* Absence of skin irritation, breakdown, and pressure injuries present in the buttocks, sacrum, and/or perineal areas at the time of enrollment; minor irritation may be acceptable at the discretion of the Study Investigator
* Willing and able to provide written informed consent or legal authorized representative is willing and able to provide written informed consent

Exclusion Criteria:

* Presence of skin irritation and/or breakdown including but not limited to IAD or pressure injuries present in the buttocks, sacrum, and/or perineal areas at the time of enrollment; minor irritation may be acceptable at the discretion of the study Investigator
* Require use of an absorbent undergarment (e.g. Depends) or catheter as the primary incontinence management strategy
* Is considered to be near death or requires hospice care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Patient exposure time following an incontinence event | Through study completion, an average of 6 months

SECONDARY OUTCOMES:
Patient satisfaction surveys | Through study completion, an average of 6 months
Staff satisfaction surveys | Through study completion, an average of 6 months
Family/patient support member surveys | Through study completion, an average of 6 months
Incidence of incontinence associated skin irritation and breakdown issues | Through study completion, an average of 6 months
Incidence of pressure injuries | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Parkview Regional Medical Center, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No